CLINICAL TRIAL: NCT05334147
Title: Anlotinib Combined With Chemotherapy for the Treatment of HER2 Negative Advanced Breast Cancer Previously Treated With Anthracyclines and Taxanes: A Multicenter, Prospective, Observational Clinical Study
Brief Title: Anlotinib Combined With Chemotherapy for the Treatment of HER2 Negative Advanced Breast Cancer
Acronym: ALOT-BC1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-SR-592
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: HER2-negative Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anlotinib in combination with chemotherapy: anlotinib12mg qd p.o. d1-14/21day/cycle；eribulin 1.4 mg/m2，d1&d8/21day/cycle；capecitabine 1000 mg/m2，bid，d1-14/21day/cycle.
- chemotherapy: eribulin 1.4 mg/m2，d1&d8/21day/cycle；capecitabine 1000 mg/m2，bid，d1-14/21day/cycle.

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of anlotinib combined with chemotherapy treatment for patients with HER2 negative advanced breast cancer previously received anthracyclines and taxanes

DETAILED DESCRIPTION:
Breast cancer is the most frequent malignancy in women worldwide. Treatments on HER2 negative breast cancer are still under exploration. Therefore, it is imperative to find a novel therapy to treat these patients.

Anlotinib is an anti-angiogenic small-molecule butyrate kinase inhibitor, and preliminary phase II study results show that anlotinib has good efficacy and tolerability in the treatment of HER-2-negative advanced breast cancer.

This study is a prospective, multicenter, observational clinical study that will collect and report anlotinib in combination with anlotinib in patients with HER2-negative advanced breast cancer treated with anthracyclines and taxanes in a real-world clinical setting Efficacy and safety data for chemotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old (calculated on the day of signing informed consent);
2. Histologically diagnosed advanced breast cancer, including inoperable locally advanced breast cancer or recurrent/metastatic breast cancer;
3. Immunohistochemical detection of HER-2 (-) or (1+), of which HER-2 (2+) must be tested by FISH and the result is negative;
4. All patients have previously underwent chemotherapy containing anthracyclines and taxanes (adjuvant, neoadjuvant or rescue therapy) , and treatment failure or disease progression received at most two chemotherapy regimens after recurrence/metastasis. HR+/HER2- breast cancer patients need to complete endocrine drug therapy;
5. Physical condition ECOG PS: 0-1;
6. There is at least 1 measurable lesion of metastasis according to RECIST 1.1;
7. The patients voluntarily joined the project and signed the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with a previous history of breast cancer were excluded, except for ipsilateral DCIS who received only local therapy ≥5 years ago; patients with a history of any other cancer (except non-melanoma skin cancer or cervical carcinoma in situ) were excluded;
3. allergic to Anlotinib;
4. Received eribulin, capecitabine treatment or anti-angiogenic drug treatment in the past;
5. Uncontrolled brain metastases (except asymptomatic, or patients with stable brain metastases receiving local treatment);
6. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 negative advanced breast cancer patients treated with anthracyclines and taxanes
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 1 year after the last patient enrolled
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause

SECONDARY OUTCOMES:
objective response rate（ORR） | up to 1 year after the last patient enrolled
  The ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)
Clinical benefit rate（CBR） | up to 1 year after the last patient enrolled
  Proportion of patients with a complete response (CR), partial response (PR), and stable disease (SD) ≥24 weeks in the best objective tumor response
overall survival（OS） | up to 1 year after the last patient enrolled
  The time from the patient's initiation of treatment to death from any cause
Incidence and Severity of adverse events | up to 1 year after the last patient enrolled
  AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Yin, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Wei Li, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Angulo AM, Morales-Vasquez F, Hortobagyi GN. Overview of resistance to systemic therapy in patients with breast cancer. Adv Exp Med Biol. 2007;608:1-22. doi: 10.1007/978-0-387-74039-3_1. PMID 17993229
- [Background] Banerjee S, Dowsett M, Ashworth A, Martin LA. Mechanisms of disease: angiogenesis and the management of breast cancer. Nat Clin Pract Oncol. 2007 Sep;4(9):536-50. doi: 10.1038/ncponc0905. PMID 17728712
- [Background] Ranpura V, Hapani S, Wu S. Treatment-related mortality with bevacizumab in cancer patients: a meta-analysis. JAMA. 2011 Feb 2;305(5):487-94. doi: 10.1001/jama.2011.51. PMID 21285426
- [Background] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Result] Hu N, Si Y, Yue J, Sun T, Wang X, Jia Z, Gao S, Li Q, Shao Y, Wang J, Luo Y, Ma F, Xu B, Yuan P. Anlotinib has good efficacy and low toxicity: a phase II study of anlotinib in pre-treated HER-2 negative metastatic breast cancer. Cancer Biol Med. 2021 Mar 12;18(3):849-59. doi: 10.20892/j.issn.2095-3941.2020.0463. PMID 33710812